CLINICAL TRIAL: NCT02357368
Title: Impact of Hormonal Contraception on HIV Acquisition and Transmission Risk
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lisa Haddad (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Lisa Haddad, Asscoiate Professor, Emory University
Organization: Emory University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00072549; 5K23HD078153-05 (NIH)
Record Dates: First submitted 2015-02-03; First posted 2015-02-06 (Estimated); Results first posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-10

CONDITIONS: HIV; Contraception
Keywords: HIV-negative
MeSH Terms: interventions — Medroxyprogesterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (4):
- Depot medroxyprogesterone acetate (DMPA) (Experimental): DMPA will be administered every 12 weeks at 150 mg by intramuscular (IM) injection at week 3 of study enrollment and repeated at week 15.
  Interventions: Drug: Depot medroxyprogesterone acetate (DMPA)
- Etonogestrel implant (Eng-Implant) (Experimental): A standard Nexplanon rod Implant will be placed at study week 3.
  Interventions: Device: Etonogestrel implant (Eng-Implant)
- Levonorgestrel intrauterine device (Lng-IUD) (Experimental): A standard Mirena IUD will be placed at study week 3.
  Interventions: Device: Levonorgestrel intrauterine device (Lng-IUD)
- ParaGard® T 380A Intrauterine Copper Contraceptive (Experimental): A standard ParaGuard IUD will be placed at study week 3.
  Interventions: Device: ParaGard® T 380A Intrauterine Copper Contraceptive

INTERVENTIONS:
Drug: Depot medroxyprogesterone acetate (DMPA) — DMPA will be administered every 12 weeks at the standard dose of 150 mg IM, beginning from week 3 of study enrollment and repeated at week 15.
  Other Names: Depo Provera
  Arms: Depot medroxyprogesterone acetate (DMPA)
Device: Etonogestrel implant (Eng-Implant) — A standard nexplanon rod implant will be placed at study week 3 by a trained clinician.
  Other Names: Nexplanon
  Arms: Etonogestrel implant (Eng-Implant)
Device: Levonorgestrel intrauterine device (Lng-IUD) — A standard Mirena IUD will be placed at study week 3 by a trained clinician.
  Other Names: Mirena
  Arms: Levonorgestrel intrauterine device (Lng-IUD)
Device: ParaGard® T 380A Intrauterine Copper Contraceptive — A standard ParaGuard IUD will be placed at study week 3 by a trained clinician.
  Other Names: ParaGuard
  Arms: ParaGard® T 380A Intrauterine Copper Contraceptive

SUMMARY:
This is a prospective cohort study focusing on HIV negative women. The investigators want to learn how the contraceptive methods of depot medroxyprogesterone acetate (DMPA), etonogestrel implant (Eng-Implant), levonorgestrel intrauterine device (Lng-IUD) and the ParaGard® T 380A Intrauterine Copper Contraceptive impact the vaginal immune environment.

DETAILED DESCRIPTION:
The three proposed aims will evaluate the effect of four contraceptive methods (depot medroxyprogesterone acetate (DMPA), etonogestrel implant (Eng-Implant), levonorgestrel intrauterine device (Lng-IUD) and ParaGard® T 380A Intrauterine Copper Contraceptive) on: (1) HIV target immune cells within the female genital mucosa; (2) markers of T-cell activation and trafficking within the female genital mucosa; and (3) secreted cytokines and chemokines within the female genital mucosa.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18-45 years
* Normal menses (22-35 day intervals) for at least 3 cycles
* Intact uterus and cervix
* Interested in to DMPA, Eng-Implant or Lng-IUD or ParaGuard
* Willing to delay initiation of hormonal contraception for up to 1 month
* Willing to use condoms or abstain from sexual intercourse for at least 48 hours before each genital tract sampling (condoms will be made available)
* Able and willing to provide informed consent, and undergo serial blood and cervicovaginal lavage (CVL) sampling
* Negative HIV screening

Exclusion Criteria:

* Pregnant within the last 3 months
* Breastfeeding
* History of loop electrosurgical excision procedure, conization, or cryosurgery within the past year
* Use of hormonal contraception or IUD in the past 6 months
* Known history of medical condition that would interfere with the conduct of the study
* Symptomatic vaginal infection or genital ulcer disease at screening
* Taking medications that interact with selected contraceptive
* Contraindications to selected contraceptive per the Centers for Disease Control and Prevention (CDC) medical eligibility criteria or judgment of clinician

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2015-02; Primary Completion 2019-10-23 (Actual); Study Completion 2019-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Haddad, MD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Grady Health System, Atlanta, Georgia
  - The Ponce de Leon Center of the Grady Health System, Atlanta, Georgia
  - Emory Clinic, Atlanta, Georgia
  - Emory University Clinical Research Network, Atlanta, Georgia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between February 2015 and follow up was completed on October 23, 2019. Participants were recruited from the Grady Family Planning Clinic within Grady Memorial Hospital, the Emory Clinic, and the Ponce de Leon Center of the Grady Health System, in Atlanta, Georgia.
Groups:
- Depot Medroxyprogesterone Acetate (DMPA): Participants receiving depot medroxyprogesterone acetate (DMPA) administered every 12 weeks at the standard dose of 150 mg intramuscular injection, beginning from Week 3 of study enrollment and repeated at Week 15
- Etonogestrel Impant (Eng-Implant): Participants receiving a standard nexplanon rod implant that was placed at study Week 3 by a trained clinician
- Levonorgestrel Intrauterine Device (Lng-IUD): Participants receiving a standard Mirena intrauterine device (IUD) that was placed at study Week 3 by a trained clinician
- ParaGard® T 380A Intrauterine Copper Contraceptive: Participants receiving a standard ParaGuard IUD that was placed at study week 3 by a trained clinician
Period: Overall Study
Arm/Group | Depot Medroxyprogesterone Acetate (DMPA) | Etonogestrel Impant (Eng-Implant) | Levonorgestrel Intrauterine Device (Lng-IUD) | ParaGard® T 380A Intrauterine Copper Contraceptive
Started | 19 | 18 | 14 | 8
Completed | 13 | 15 | 13 | 5
Not Completed | 6 | 3 | 1 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Pregnancy | 3 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Depot Medroxyprogesterone Acetate (DMPA): Participants receiving DMPA administered every 12 weeks at the standard dose of 150 mg intramuscular injection, beginning from Week 3 of study enrollment and repeated at Week 15
- Levonorgestrel Intrauterine Device (Lng-IUD): Participants receiving a standard Mirena IUD that was placed at study Week 3 by a trained clinician
- Total: Total of all reporting groups
Arm/Group | Depot Medroxyprogesterone Acetate (DMPA) | Etonogestrel Impant (Eng-Implant) | Levonorgestrel Intrauterine Device (Lng-IUD) | ParaGard® T 380A Intrauterine Copper Contraceptive | Total
Number analyzed (Participants) | 19 | 18 | 14 | 8 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 18 | 14 | 8 | 59
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Continuous age is not available for the ParaGard® T 380A Intrauterine Copper Contraceptive study arm. This group was added late in the study and the study procedures differed slightly from the initial three study arms.
  years
    number analyzed (Participants) | 19 | 18 | 14 | 0 | 51
    (all) | 34.1 (7.8) | 27.7 (7.2) | 31.1 (7.9) |  | 31.0 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 14 | 8 | 59
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity is not available for the ParaGard® T 380A Intrauterine Copper Contraceptive study arm. This group was added late in the study and the study procedures differed slightly from the initial three study arms.
  Participants
    number analyzed (Participants) | 19 | 18 | 14 | 0 | 51
    Hispanic or Latino | 1 | 1 | 0 |  | 2
    Not Hispanic or Latino | 18 | 17 | 14 |  | 49
    Unknown or Not Reported | 0 | 0 | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race is not available for the ParaGard® T 380A Intrauterine Copper Contraceptive study arm. This group was added late in the study and the study procedures differed slightly from the initial three study arms.
  Participants
    number analyzed (Participants) | 19 | 18 | 14 | 0 | 51
    American Indian or Alaska Native | 0 | 0 | 0 |  | 0
    Asian | 0 | 0 | 0 |  | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 |  | 0
    Black or African American | 18 | 15 | 7 |  | 40
    White | 1 | 2 | 7 |  | 10
    More than one race | 0 | 1 | 0 |  | 1
    Unknown or Not Reported | 0 | 0 | 0 |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 18 | 14 | 8 | 59

OUTCOME MEASURES:

1. Primary Outcome: Percent of HIV Target Immune Cells Within Female Genital Mucosa and Blood
Description: Following exposure to HIV, initial infection occurs at the genital mucosa and may involve complex interactions between a number of HIV target immune cells. HIV often uses C-C Chemokine Receptor Type 5 (CCR5) for entrance into target immune cells, causing infection of the cell. The amount of CCR5 expressing macrophages is associated with HIV infection. Cluster of differentiation 4 (CD4) T Cells are targeted and infected by HIV and CD4 percentages are used to assess immune status. CD4 counts vary by individuals and generally decrease with HIV infection.
Time Frame: Week 1, Week 17
Measure: Mean (Standard Deviation); unit: percentage of HIV target immune cells
Arm/Group | Depot Medroxyprogesterone Acetate (DMPA) | Etonogestrel Impant (Eng-Implant) | Levonorgestrel Intrauterine Device (Lng-IUD) | ParaGard® T 380A Intrauterine Copper Contraceptive
Number analyzed (Participants) | 19 | 18 | 14 | 8
percentage of HIV target immune cells
  CCR5+ CD4 T-cells Cervicovaginal Lavage (CVL) Week 1 | 26.6 (22.3) | 22.8 (20.5) | 16.9 (16.4) | 22.4 (20.3)
  CCR5+ CD4 T-cells CVL Week 17 | 39.2 (27.6) | 32.2 (21.1) | 23.3 (20.6) | 15.3 (8.1)
  CCR5+ CD4 T-cells Peripheral Blood Mononuclear Cell (PBMC) Week 1 | 4.1 (2.9) | 3.9 (2.5) | 2.9 (1.7) | 8.3 (2.9)
  CCR5+ CD4 T-cells PBMC Week 17 | 5.7 (3.5) | 4.2 (2.7) | 2.6 (1.4) | 7.5 (1.6)
  CD4% CVL Week 1 | 47.2 (17.5) | 48.7 (16.7) | 54.0 (20.5) | 63.4 (11.2)
  CD4% CVL Week 17 | 47.4 (18.2) | 47.0 (16.3) | 48.8 (23.5) | 47.5 (22.7)
  CD4% PBMC Week 1 | 65.6 (10.6) | 67.4 (8.0) | 65.7 (9.4) | 73.3 (4.9)
  CD4% PBMC Week 17 | 63.9 (10.1) | 67.5 (9.4) | 63.4 (10.8) | 71.1 (13.7)

2. Primary Outcome: Ratio of CD4/Cluster of Differentiation 8 (CD8) T-Cells Within Female Genital Mucosa and Blood
Description: CD4/CD8 ratios above 1 indicate a strong immune system while lower ratios indicate a viral infection.
Time Frame: Week 1, Week 17
Measure: Mean (Standard Deviation); unit: CD4/CD8
Arm/Group | Depot Medroxyprogesterone Acetate (DMPA) | Etonogestrel Impant (Eng-Implant) | Levonorgestrel Intrauterine Device (Lng-IUD) | ParaGard® T 380A Intrauterine Copper Contraceptive
Number analyzed (Participants) | 19 | 18 | 14 | 8
CD4/CD8
  CD4/CD8 Ratio Cervicovaginal Lavage (CVL) Week 1 | 2.4 (2.5) | 2.6 (1.8) | 2.9 (3.0) | 3.9 (3.0)
  CD4/CD8 Ratio CVL Week 17 | 2.6 (2.7) | 2.3 (2.0) | 2.3 (2.1) | 4.9 (6.5)
  CD4/CD8 Ratio Peripheral Blood Mononuclear Cell (PBMC) Week 1 | 4.3 (8.8) | 3.1 (1.7) | 2.9 (1.5) | 4.7 (2.0)
  CD4/CD8 Ratio PBMC Week 17 | 2.6 (1.3) | 3.3 (2.5) | 2.5 (1.2) | 5.4 (2.1)

3. Primary Outcome: Percent of Markers of T-cell Activation and Trafficking Within the Female Genital Mucosa and Blood
Description: T cell activation correlates with HIV infection progression and this study seeks to gain better understanding of these underlying mechanisms by assessment of HIV target cells. Changes in cluster of differentiation 38 (CD38) expression are indicators of HIV disease progression with increases seen in CD38+ when a chronic HIV infection is progressing. Human leukocyte antigen-antigen D related (HLA-DR)+ expression appears to be involved in HIV proliferation.
Time Frame: Week 1, Week 17
Population: This analysis includes participants with samples that were able to be analyzed. Missing values are due to the inability to quantify the outcomes due to low cell counts when looking at the percent + of few cells for those samples.
Measure: Mean (Standard Deviation); unit: percentage of T cell activation markers
Arm/Group | Depot Medroxyprogesterone Acetate (DMPA) | Etonogestrel Impant (Eng-Implant) | Levonorgestrel Intrauterine Device (Lng-IUD) | ParaGard® T 380A Intrauterine Copper Contraceptive
Number analyzed (Participants) | 19 | 18 | 14 | 8
percentage of T cell activation markers
  CD38+ CD4 T-cells Cervicovaginal Lavage (CVL) Week 1 | 36.7 (18.4) | 36.9 (17.6) | 32.6 (11.6) | 23.2 (22.4)
  CD38+ CD4 T-cells CVL Week 17 | 35.9 (18.6) | 41.7 (14.8) | 44.0 (15.4) | 45.5 (21.4)
  CD38+ CD4 T-cells Peripheral Blood Mononuclear Cell (PBMC) Week 1 | 17.1 (7.3) | 17.6 (10.1) | 17.0 (9.0) | 25.2 (10.4)
  CD38+ CD4 T-cells PBMC Week 17 | 17.7 (6.9) | 17.6 (8.4) | 17.2 (7.0) | 36.3 (25.0)
  HLA-DR+ CD4 T-cells CVL Week 1 | 25.0 (18.3) | 26.9 (22.8) | 15.4 (10.4) | 8.7 (6.1)
  HLA-DR+ CD4 T-cells CVL Week 17 | 21.2 (16.6) | 17.8 (13.8) | 11.4 (6.9) | 21.1 (19.1)
  HLA-DR+ CD4 T-cells PBMC Week 1 | 4.8 (3.4) | 3.0 (1.5) | 3.3 (2.1) | 3.4 (1.4)
  HLA-DR+ CD4 T-cells PBMC Week 17 | 4.4 (2.9) | 2.3 (0.9) | 3.6 (6.2) | 2.5 (1.6)
  CD38+ Target (CCR5+ CD4+) T cells CVL Week 1: number analyzed (Participants) | 17 | 17 | 14 | 8
  CD38+ Target (CCR5+ CD4+) T cells CVL Week 1 | 62.5 (20.6) | 64.5 (26.9) | 66.2 (18.4) | 12.7 (13.9)
  CD38+ Target (CCR5+ CD4+) T cells CVL Week 17: number analyzed (Participants) | 17 | 17 | 14 | 8
  CD38+ Target (CCR5+ CD4+) T cells CVL Week 17 | 52.5 (20.7) | 61.6 (14.7) | 70.8 (18.9) | 42.4 (29.4)
  CD38+ Target (CCR5+ CD4+) T cells PBMC Week 1 | 22.7 (8.6) | 26.0 (12.8) | 28.2 (10.6) | 18.6 (12.6)
  CD38+ Target (CCR5+ CD4+) T cells PBMC Week 17 | 24.1 (9.2) | 29.6 (12.1) | 31.7 (9.7) | 30.9 (20.3)
  HLA-DR+ Target (CCR5+ CD4+) T cells CVL Week 1: number analyzed (Participants) | 17 | 17 | 14 | 8
  HLA-DR+ Target (CCR5+ CD4+) T cells CVL Week 1 | 30.7 (21.6) | 41.3 (24.8) | 28.2 (16.3) | 20.1 (12.9)
  HLA-DR+ Target (CCR5+ CD4+) T cells CVL Week 17: number analyzed (Participants) | 17 | 17 | 14 | 8
  HLA-DR+ Target (CCR5+ CD4+) T cells CVL Week 17 | 30.0 (17.6) | 25.5 (17.9) | 17.6 (11.9) | 26.5 (18.7)
  HLA-DR+ Target (CCR5+ CD4+) T cells PBMC Week 1 | 24.4 (10.4) | 22.6 (7.4) | 28.3 (10.1) | 16.5 (9.9)
  HLA-DR+ Target (CCR5+ CD4+) T cells PBMC Week 17 | 23.2 (10.4) | 21.6 (7.6) | 25.5 (11.6) | 10.1 (7.3)

4. Primary Outcome: Concentration Levels of Secreted Cytokines and Chemokines Within the Female Genital Mucosa and Blood
Description: The concentration levels of interleukin 1 (IL-1) family cytokines and interferon gamma-induced protein 10 (IP-10) chemokines were determined using multiplex Luminex® assays combined with a customized multi-analytical panel of 22 human cytokines and chemokines. IL-1 and IP-10 have been found to influence recruitment of HIV target cells to the female reproductive tract and this study is examining changes in IL-1 and PI-10 to gain further understanding of these mechanisms.
Time Frame: Week 1, Week 17
Population: The ParaGard® T 380A Intrauterine Copper Contraceptive study arm was added late in the study the study procedures differed slightly from the initial three study arms. Funding to add this study arm covered the evaluation of the clinical study activities and cellular markers and there was not funding for analysis of cytokines and chemokines.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Depot Medroxyprogesterone Acetate (DMPA) | Etonogestrel Impant (Eng-Implant) | Levonorgestrel Intrauterine Device (Lng-IUD) | ParaGard® T 380A Intrauterine Copper Contraceptive
Number analyzed (Participants) | 19 | 18 | 14 | 0
pg/mL
  IP-10 Cervicovaginal Lavage (CVL) Week 1 | 689.8 (1052.5) | 2551.1 (2936.2) | 1100.2 (1974.1) |
  IP-10 CVL Week 17 | 445.8 (996.1) | 2417.6 (3667.7) | 1241.5 (1088.5) |
  IP-10 Peripheral Blood Mononuclear Cell (PBMC) Week 1 | 3298.5 (2066.1) | 4107.3 (1455.4) | 204.4 (83.4) |
  IP-10 PBMC Week 17 | 3114.4 (1843.8) | 3954.3 (1617.0) | 209.6 (75.7) |
  IL-1a CVL Week 1 | 752.2 (1616.8) | 1640.2 (2051.6) | 256.4 (413.1) |
  IL-1a CVL Week 17 | 550.7 (695.8) | 2120.6 (2569.5) | 184.7 (251.0) |
  IL-1a PBMC Week 1 | 58.5 (154.2) | 156.2 (233.2) | 54.6 (87.7) |
  IL-1a PBMC Week 17 | 47.8 (118.2) | 144.1 (235.9) | 65.1 (78.5) |
  IL-1b CVL Week 1 | 32.9 (50.3) | 583.4 (1569.9) | 43.9 (91.3) |
  IL-1b CVL Week 17 | 21.1 (42.0) | 485.8 (971.9) | 37.1 (30.8) |
  IL-1b PBMC Week 1 | 20.0 (11.2) | 51.4 (73.2) | 4.2 (2.3) |
  IL-1b PBMC Week 17 | 20.8 (10.8) | 46.5 (58.1) | 4.3 (1.9) |

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected from the time of giving consent to participate through Study Visit 4 (Week 17).
Arm/Group | Depot Medroxyprogesterone Acetate (DMPA) | Etonogestrel Impant (Eng-Implant) | Levonorgestrel Intrauterine Device (Lng-IUD) | ParaGard® T 380A Intrauterine Copper Contraceptive
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/18 | 0/14 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18 | 0/14 | 0/8
Other Adverse Events (participants affected / at risk) | 1/19 | 0/18 | 1/14 | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Depot Medroxyprogesterone Acetate (DMPA) (N=19) | Etonogestrel Impant (Eng-Implant) (N=18) | Levonorgestrel Intrauterine Device (Lng-IUD) (N=14) | ParaGard® T 380A Intrauterine Copper Contraceptive (N=8)
Extended spotting 7 days before start of menstrual cycle (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Extended menstrual bleeding with blood clots (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Heavy irregular menstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/68/NCT02357368/Prot_SAP_000.pdf
  • Informed Consent Form (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/68/NCT02357368/ICF_001.pdf